CLINICAL TRIAL: NCT05035888
Title: Prophylactic Norepinephrine and Phenylephrine Boluses for Postspinal Anesthesia Hypotension in Patients Undergoing Caesarean Section: A Randomized Sequential Allocation Dose-finding Study.
Brief Title: Prophylactic Norepinephrine and Phenylephrine Boluses for Postspinal Anesthesia Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2021-6
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-09

CONDITIONS: Adverse Effect
Keywords: Norepinephrine; Phenylephrine; Postspinal anesthesia hypotension; Cesarean section
MeSH Terms: interventions — Phenylephrine; Vasoconstrictor Agents; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine group (Active Comparator): Prophylactic phenylephrine bolus simultaneous with spinal anesthesia
  Interventions: Drug: Phenylephrine
- Norepinephrine group (Experimental): Prophylactic norepinephrine bolus simultaneous with spinal anesthesia
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — An initial prophylactic bolus dose of phenylephrine (37.5μg) simultaneous with spinal anesthesia. If the patient did not respond adequately to the current dose (SBP decreased to < 80% of baseline), the dose was considered to have failed and the subsequent dose for the following patient was increased to the next higher dose level. The dose administered to subsequent patients varied by increments or decrements of 12.5 μg according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Vasopressors
  Arms: Phenylephrine group
Drug: Norepinephrine — An initial prophylactic bolus dose of norepinephrine (3μg) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 1 μg according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Vasopressors
  Arms: Norepinephrine group

SUMMARY:
The purpose of this study is to investigate the potency between prophylactic norepinephrine and phenylephrine boluses for postspinal anesthesia hypotension in patients undergoing caesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Vasopressor has been highly recommended for routine prevention and/or treatment of post-spinal anesthesia hypotension. As a potential substitute drug for phenylephrine, norepinephrine has gradually been used in parturients undergoing cesarean section. There's some evidence that prophylactic infusion of norepinephrine could effectively reduce the incidence of post-spinal anesthesia hypotension in parturients undergoing cesarean section. However, few studies had been indicated the ED50 (prevent postspinal hypotension in 50% of patients) and ED90 of prophylactic norepinephrine bolus and its potency compared to phenylephrine for postspinal anesthesia hypotension in patients undergoing caesarean section. The purpose of this study is to investigate the potency between prophylactic norepinephrine and phenylephrine boluses for postspinal anesthesia hypotension in patients undergoing caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥180 mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
The dose that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) and 90% (ED90) of patients | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China